CLINICAL TRIAL: NCT07125612
Title: Impact of Perioperative Allogeneic Red Blood Cell Transfusion on Postoperative Myocardial Injury After Liver Resection
Status: Completed | Type: Observational
Sponsor: Hao Li (Other)
Responsible Party: Sponsor-Investigator, Hao Li, Professor, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: ChinaPLAGH_transfusion
Record Dates: First submitted 2025-08-09; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Myocardial Injury; Acuter Kidney Injury
Keywords: perioperative allogeneic red blood cell transfusion; elderly surgical patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aimed to explore the influence of ABT on the incidence of MINS, AKI, and overall prognosis among advanced-age HCC patients who underwent hepatectomy

ELIGIBILITY:
Inclusion Criteria:

Patients over 65 years with HCC undergoing elective surgery between January 2016 and December 2018

Exclusion Criteria:

ASA grade V requiring repeat surgery within 1 week losing to follow-up and/or those with >5% missing data

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: age ≥65 years old patients
Sampling Method: Non-Probability Sample
Enrollment: 487 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
the incidence of MINS within postoperative 30 days | postoperative day 1-30

SECONDARY OUTCOMES:
overall survival (OS) | postoperative day 1-30
  the time from the date of surgery to the date of death
postoperative 7-day AKI | postoperative day 1-7

IPD SHARING:
Plan to Share IPD: No